CLINICAL TRIAL: NCT01403896
Title: A Pilot Study To Design a Clinical Trial That Will Compare the Ability of Plerixafor Alone Versus Plerixafor Plus G-CSF To Generate a Bone Marrow Versus Blood Transplant Product In Normal Healthy Adults
Brief Title: Healthy Donor Study II - Comparing Plerixafor With G-CSF and Plerixafor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Couban (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Stephen Couban, Hematologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC001
Record Dates: First submitted 2011-07-14; First posted 2011-07-27 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Malignant Lymphoma, Stem Cell Type
Keywords: Hematopoietic Stem Cell Transplantation; Plerixafor; Healthy Donors; Stem Cell Graft
MeSH Terms: conditions — Lymphoma | interventions — plerixafor; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plerixafor Group (Active Comparator)
  Interventions: Drug: Plerixafor (Mozobil)
- Plerixafor + G-CSF group (Experimental)
  Interventions: Drug: Plerixafor + G-CSF

INTERVENTIONS:
Drug: Plerixafor (Mozobil) — They will receive Plerixafor (240 µg/kg/day subcutaneously for 1 dose) on Day 0 at 8 am
  Other Names: Mozobil; AMD 3100
  Arms: Plerixafor Group
Drug: Plerixafor + G-CSF — They will receive G-CSF (5 µg/kg/day) for 4 days (Days -4,-3,-2,-1 at 8 am) followed by Plerixafor (240 µg/kg/day subcutaneously for 1 dose) on Day 0 at 8 am
  Other Names: Mozobil; AMD 3100; Neupogen
  Arms: Plerixafor + G-CSF group

SUMMARY:
Stem cells can be transplanted from a healthy donor to a patient to combat blood cancers and other disorders. This process is called stem cell transplantation. Stem cells normally live in the bone marrow. A bone marrow transplantation (BMT) is when the bone marrow is directly transplanted into a patient. However, stem cells can also be stimulated to move from the bone marrow to the blood where they can be collected, a process is called mobilization. When these stem cells are transplanted it is called peripheral blood stem cell transplantation (PBSCT). Both stem cell sources are used for different reasons, but PBSCT is much more common.

There is considerable debate as to which stem cell source, BMT or PBSCT, is optimal. There are differences between the two sources in important transplant outcomes. The stem cell product that is transplanted, also called the stem cell graft, contains more than just stem cells. Results from studies suggest that the variation in the cells with grafts may account for the variation in outcomes. Preliminary data from a recent study conducted by the Canadian Blood and Bone Marrow Transplant Group has associated relative frequencies of particular cell populations with leukemic relapse and another important outcome called graft versus host disease (GVHD). While the later essentially equates to a failed transplant, the former is the most common and devastating complication of stem cell transplantation.

The only drug used to mobilize stem cells into the blood of health donors for collection is G-CSF. However there is a new mobilization drug recently approved called plerixafor. This drug is able to mobilize stem cells when G-CSF has failed and pre-clinical studies suggest that it may produce a superior stem cell graft to G-CSF alone. There is little information available, besides safety and efficacy data, about the effects that plerixafor has on the stem cell graft of normal healthy donors.

This study will compare the stem cell graft in normal healthy donors following plerixafor mobilization versus plerixafor and G-CSF mobilization. Specifically, they will look at the cell populations that have been previously correlated with important transplantation outcomes like relapse and GVHD. The investigators suspect that the stem cell graft mobilized by plerixafor and G-CSF will provide a superior graft to that mobilized by plerixafor alone.

DETAILED DESCRIPTION:
Background:

Stem cell transplantation (SCT) involves transfusing stem cells collected from 3 potential sources: bone marrow, peripheral blood, or umbilical cord. There are 2 major types of transplantation. Autologous SCT involves transplanting the patients own stem cells, while allogeneic transplantation involves transplanting stem cells from someone else. Whatever the source, the transplanted stem cell product is called the graft. Currently, the most common source is peripheral blood, However, there is considerably debate as to the optimal stem cell source because different sources have been associated with different transplant outcomes. One key outcome is graft versus host disease (GVHD). This is the most common complication of SCT and contributes significantly to transplant morbidity and mortality, as well as relapse.

Stem cells normally populate the bone marrow. Drugs are used to encourage stem cells to go into the peripheral blood, a process call mobilization. In the peripheral blood stem cells can be collected and subsequently transplanted. In Canada, the only drug used to mobilize stem cells from donors is filgrastim, a form of granulocyte colony stimulating factor (G-CSF). Although well tolerated, there are some shortcomings to this agent and there is clearly room to improve in terms of the donor experience and providing the optimal stem cell graft.

A soon to be completed study conducted by the Canadian Blood and Bone Marrow Transplant Group (CBMTG), called CBMTG 0601, is evaluating the best stem cell source. The study is aimed to compare the outcomes between allogeneic transplant patients who receive either G-CSF stimulated bone marrow or peripheral blood. This will be a seminal study that should provide valuable information as to the optimal stem cell source in allogeneic SCT. Early results suggest that the investigators may be able to predict important SCT outcomes, such as transplant related mortality, relapse or graft versus host disease, by looking at cell populations in the graft.

Plerixafor is a new mobilization agent that is approved for use in combination with neupogen in myeloma and relapsed lymphoma who are undergoing an autologous SCT. Following numerous publications on the safety and dosing of plerixafor, there were 2 pivotal high quality studies performed in this patient population. The results of this study lead to FDA approval, and Health Canada approval is close. Plerixafor may be a clinically superior mobilizing agent to Neupogen. More importantly though, it has a formidable safety profile and arguably superior in this respect. There has also been a case report and a trial demonstrating both the safety and efficacy of plerixafor in healthy donors as well. Finally, preclinical work suggests that plerixafor mobilization may yield a superior graft. Taken together, this work supports the notion that plerixafor may be a superior mobilization agent over neupogen.

Rationale:

Considering the shortcomings of neupogen and the demonstrated potential of plerixafor in trials with autologous SCT patients, it would be logical to further investigate the efficacy of plerixafor in normal healthy donors for allogeneic SCT. The investigators can confidently state that plerixafor is safe. Furthermore, plerixafor can mobilize myeloma and lymphoma patients who have failed neupogen mobilization. However, although suggested in preclinical data, there is no firm evidence to suggest that plerixafor mobilization provides a superior stem cell graft. The investigators will administer either plerixafor or plerixafor and neupogen then compare the cell populations in both peripheral blood and bone marrow..

Importance:

The use of SCT has steadily increased in the last 20 years. This has especially increased since using neupogen to mobilize stem cells thereby making transplants easier. Now that there is a new agent available that is likely safer and perhaps more efficacious, its use may improve both donor experience and patient outcomes. If plerixafor grafts consist of cell populations that are associated with superior transplant outcomes as determined in CBMTG 0601, then it will likely be used in an upcoming larger clinical trial comparing neupogen and plerixafor in normal healthy donors.

Objectives:

Our primary objective is to determine the best timing for harvesting stem cells from normal donors given plerixafor with or without neupogen. A secondary objective is to evaluate and compare the change over time after plerixafor with or without neupogen administration on the population of cells in the graft predicted to give superior transplant outcomes. The other secondary objective is to evaluate and compare the change over time after plerixafor with or without neupogen administration on the concentration of cells in the PB and BM of normal donors predicted to give GVHD or relapse. The investigators hypothesise that plerixafor with neupogen will provide a graft with increased cell populations associated with superior SCT outcomes.

ELIGIBILITY:
The inclusion and exclusion criteria are designed to reflect those that are used in practice to choose appropriate normal healthy donors for allogeneic stem cell transplantation.

Inclusion Criteria:

* Male or female between the ages of 18 and 30
* Unable or unwilling to give written informed consent
* No history of cardiac, pulmonary, liver or renal disease
* Normal CBC, creatinine, liver enzymes, bilirubin, INR and PTT

Exclusion Criteria:

* Allergy to G or to E.coli-derived agents
* Allergy to "caine" type anesthetics
* Pregnancy or breast feeding
* BMI greater than 25 to avoid difficulty with the number of bone marrows performed
* Skin conditions, autoimmune disease, sickle cell disease or splenomegaly to avoid rare side effects of G-CSF
* Any subject, who in the opinion of the investigator, should not participate in this study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The frequency of CD34+ and CD34+CD38- cells at different time points as compared to baseline. | Day -1, 0, +1
  The frequency of CD34+ and CD34+CD38- cells in a graft has been show to be an excellent measure of hematopoietic engrafting potential.

SECONDARY OUTCOMES:
The frequency of CD56bright NK cells, CD4+ central memory T-cells, perforin+ CD8+ T-cells and CD19+ CD27-TLR9+ B-cells at different time points as compared to baseline. | Day -1, 0, +1
  Relative frequencies of CD56bright NK cells, CD4+ central memory T-cells, perforin+ CD8+ T-cells, and CD19+ CD27-TLR9+ B-cells has been associated with GVHD.
The frequency of CD56bright NK cells at different time points as compared to baseline | Day -1, 0, +1
  A high frequency of CD56bright NK cells in the stem cell graft has been associated with low leukemia relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Couban, Principal Investigator — CDHA
Locations (1):
- Capital Health District Authority, Halifax, Nova Scotia, Canada